CLINICAL TRIAL: NCT02100254
Title: CRC Screening Thoughts and Feelings: Increasing Engagement of African Americans
Brief Title: Narrative or Fact-Based Videos in Increasing Colorectal Cancer Screenings in African American Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I 159309; NCI-2013-01707 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 159309 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2014-03-12; First posted 2014-03-31 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer; Healthy, no Evidence of Disease
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (personal narrative) (Experimental): Participants view videos with information about CRC and screening delivered by personal narrative.
  Interventions: Behavioral: behavioral intervention
- Arm II (fact-based message) (Active Comparator): Participants view videos with information about CRC and screening delivered by informative fact-based message.
  Interventions: Behavioral: behavioral intervention

INTERVENTIONS:
Behavioral: behavioral intervention — View personal narrative informational video
  Other Names: Behavior Conditioning Therapy; Behavior Therapy; Behavioral Modification; Behavioral Therapy; Behavioral Treatment
  Arms: Arm I (personal narrative)
Behavioral: behavioral intervention — View fact-based informational video
  Other Names: Behavior Conditioning Therapy; Behavior Therapy; Behavioral Modification; Behavioral Therapy; Behavioral Treatment
  Arms: Arm II (fact-based message)

SUMMARY:
This randomized clinical trial studies narrative or fact-based videos in increasing colorectal cancer screenings in African American communities. Informational videotapes may help increase the number of participants who engage in colonoscopy screenings. It is not yet known whether narrative videos may be more effective than fact-based videos in increasing colorectal cancer screenings.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess both individual and environmental factors that guide decisions and behaviors to engage or not engage in colonoscopy screenings for African Americans in the two communities.

II. Using a Community-Based Participatory Research (CBPR) approach, develop and pilot a peer-led, narrative-based colorectal cancer behavioral intervention for increasing colonoscopy screening behaviors in African Americans.

III. Examine the efficacy of a narrative communication-style group intervention compared to a didactic intervention to influence African Americans' engagement in colorectal cancer screening, including examining the degree to which the community interventions impact cognitive and affective decision making factors about health care seeking.

IV. Examine and explore contextual factors that may influence the process of behavior change to better understand colorectal cancer (CRC) screening and health care seeking behaviors.

OUTLINE: Program locations are randomized to 1 of 2 arms.

ARM I: Participants view videos with information about CRC and screening delivered by personal narrative.

ARM II: Participants view videos with information about CRC and screening delivered by informative fact-based message.

After completion of study, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants in each component (focus groups, surveys and educational programs) will be 18 years of age and over; these men and women are generally healthy, ambulatory and able to participate in events in their community; no women, men, or children of any ethnic or social background will be excluded from the educational program
* EDUCATIONAL INTERVENTION:
* Currently non-adherent to colorectal cancer screening
* Self-identify as African American
* Are 50 years of age or older
* Have the ability to provide informed consent in English
* FOLLOW-UP ASSESSMENTS:
* Must be non-adherent for CRC screening at the time of the educational program
* Have telephone service (mobile or landline), to participate in the follow up interviews
* Agree to providing consent for release/review of their medical record

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1310 (Actual)
Dates: Start 2009-10-01; Primary Completion 2016-09-23 (Actual); Study Completion 2017-09-23 (Actual)

PRIMARY OUTCOMES:
Change in likelihood of CRC screening in previously unscreened subjects | Baseline to 6 months post-presentation
  A change score (post-presentation minus pre-presentation) will be created and summarized. In addition, the change score will be further dichotomized (e.g. increase versus no increase in the likelihood of screening) and the percent of those who experienced an increased likelihood, denoted by pi, will be computed. A corresponding 95% confidence interval will be calculated. To test for differences in variables collected pre- and post-presentation, generalized mixed linear models will be used. Testing will be done at the 0.0.5 nominal significance level and using the approximate t-test method.

SECONDARY OUTCOMES:
Number of negative affective responses to CRC screening per Affective Associations and Affectively-Based Risk surveys | Post-presentation up to 6 months
  A linear mixed model (LMM) will be employed and implemented in the SAS program MIXED.
Number of positive cognitive responses to CRC screening per Cognitively-Based Perceived Risk survey | Post-presentation up to 6 months
  An LMM will be employed and implemented in the SAS program MIXED.
Number of participants who had or scheduled colonoscopy | Up to 6 months
  A generalized linear model with a logit link function will be used.
Number of participants who performed the fecal occult blood test (FOBT)/fecal immunohistochemistry test (FIT) | Up to 6 months
  A generalized linear model with a logit link function will be used.
Number of participants who discussed CRC screening with their primary care physician | Up to 6 months
  A generalized linear model with a logit link function will be used.
Influential factors in behavior changes, assessed using qualitative analyses of text from participant interviews, including affective associations with the program, participants' cognitive-affective influences, and predisposing influences | Baseline to 1 week post-presentation & 6-months
  Qualitative text from a text analysis program will be funneled into categories using the PEN-3 and analyzed according to the categories' role and influence. Findings will be examined in comparison to quantitative data regarding the content of the intervention.
Influential factors in behavior changes, assessed using qualitative analyses of text from participant interviews, including affective associations with the program, participants' cognitive-affective influences, and predisposing influences | 1 week post-presentation to 6 months
  Qualitative text from a text analysis program will be funneled into categories using the PEN-3 and analyzed according to the categories' role and influence. Findings will be examined in comparison to quantitative data regarding the content of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Erwin, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai School of Medicine, New York, New York

REFERENCES:
- [Derived] Kiviniemi MT, Klasko-Foster LB, Erwin DO, Jandorf L. Decision-making and socioeconomic disparities in colonoscopy screening in African Americans. Health Psychol. 2018 May;37(5):481-490. doi: 10.1037/hea0000603. Epub 2018 Mar 29. PMID 29595298